CLINICAL TRIAL: NCT00005559
Title: Statistical Basis for Hemochromatosis Screening
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5104; R15HL058203 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-03

CONDITIONS: Blood Disease; Hemochromatosis
MeSH Terms: conditions — Hematologic Diseases; Hemochromatosis

SUMMARY:
To determine optimal values for transferrin saturation for use in population screening for hereditary hemochromatosis.

DETAILED DESCRIPTION:
BACKGROUND:

Once considered to be a rare disorder, hemochromatosis is now recognized to be one of the most common autosomal recessive disorders in white populations. Substantial morbidity and mortality may result from untreated hemochromatosis; thus, early detection and treatment are essential. The Centers for Disease Control and Prevention and the College of American Pathologists now recommend regular screening for hereditary hemochromatosis. Transferrin saturation is regarded as the best single screening test for the detection of individuals at risk for the disorder.

DESIGN NARRATIVE:

Statistical mixture modeling was used to develop guidelines for hemochromatosis screening regimes and to determine the frequency of the gene for hemochromatosis. The research was designed to provide a statistical foundation for the analysis of population transferrin saturations to assist in development of optimal screening regimens for hemochromatosis. To determine potential screening thresholds, probability methods were applied to data from the third National Health and Nutrition Examination Survey (NHANES III), a cross-sectional probability sample weighted to represent the U.S. population. Statistical mixture modeling was used to determine potential transferrin saturation screening thresholds to identify individuals for repeat testing and possible further evaluation. The actual sensitivity and specificity of these screening thresholds was then assessed using data from a separate demonstration project, "Cost effective Hemochromatosis Survey in Primary Care", designed to identify individuals with hemochromatosis. In addition, the gene frequency for hemochromatosis for whites and ethnic subgroups was also determined by analysis of transferrin saturation data from NHANES III.

The study has two specific aims, as follow: (1) to develop guidelines for the use of transferrin saturation and related tests in detection of individuals at risk for hemochromatosis, and (2) to determine the frequency of the gene for hemochromatosis in the United States by statistical mixture modeling of population transferrin saturation data from NHANES III. Providing the statistical foundation for the analysis of transferrin saturations should facilitate development of optimal, cost-effective screening regimens for identification of individuals requiring further evaluation for hemochromatosis.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Mc Laren — Moorhead State University

REFERENCES:
- [Background] Adams PC, Kertesz AE, McLaren CE, Barr R, Bamford A, Chakrabarti S. Population screening for hemochromatosis: a comparison of unbound iron-binding capacity, transferrin saturation, and C282Y genotyping in 5,211 voluntary blood donors. Hepatology. 2000 May;31(5):1160-4. doi: 10.1053/he.2000.6984. PMID 10796893
- [Background] McLaren CE, Li KT, Gordeuk VR, Hasselblad V, McLaren GD. Relationship between transferrin saturation and iron stores in the African American and US Caucasian populations: analysis of data from the third National Health and Nutrition Examination Survey. Blood. 2001 Oct 15;98(8):2345-51. doi: 10.1182/blood.v98.8.2345. PMID 11588029